## **AUREA**

Phase II, multicenter, non-randomized, single-arm, open-label trial of atezolizumab in combination of split-doses of gemcitabine plus cisplatin in patients with locally advanced or metastatic urothelial carcinoma

#### STATISTICAL ANALYSIS REPORT

**JULY 2023** 

Done by: MFAR CLINICAL RESEARCH S.L





# 1. TABLE OF CONTENTS

| 2. | Study design | 4 |
|---|---|---|
| 3. | Screening failure | 5 |
| 4. | Study populations | 7 |
| | 4.1. Intent-To-Treat | 7 |
| | 4.2. Per protocol | 8 |
| | 4.3. Safety population | 9 |
| 5. | Basal information | 10 |
| | 5.1. Non-cisplatin eligible | 10 |
| | 5.2. Cancer history | 12 |
| | 5.2.1. Primary cancer | 12 |
| | 5.3. Demographic data | 20 |
| | 5.4. Comorbidities and concomitant medication | 22 |
| | 5.5. Hematology and coagulation | 23 |
| | 5.6. Biochemistry, serology and thyroid function | 24 |
| | 5.7. Other determinations | 26 |
| 6. | Treatment compliance | 27 |
| | 6.1. Initial phase: Combined treatment (C1-C6) atezolizumab, cisplatin and | |
| | gemcitabine | 27 |
| | 6.2. Monotherapy phase: Adherence to atezolizumab and entire treatment | 36 |
| 7. | End of treatment | 40 |
| 8. | Efficacy analysis | 45 |
| | 8.1. Primary objective | 45 |
| | 8.1.1. Overall response rate (ORR) | 45 |
| | 8.1.1.1. ORR vs Age>70 | 47 |
| | 8.1.1.2. ORR vs Renal Impairment | 48 |
| | 8.1.1.3. ORR vs ECOG 2 | 49 |
| | 8.1.1.4. ORR vs HEMOGLOBIN | 50 |
| | 8.1.1.5. ORR vs LIVER METASTASIS | 51 |
| | 8.2. Secondary objectives | 52 |
| | 8.2.1. Time to response | 52 |
| | 8.2.2. Duration of response | 52 |
| | 8.2.3. Clinical benefit rate | 54 |
| | 8.2.4. Follow-up time | 54 |
| | 8.2.5. PFS | 55 |
| | 8.2.5.1. PFS vs Age>70 | 57 |
| | 8.2.5.2. PFS vs Renal Impairment | 58 |

| 8.2.5.3. PFS vs ECOG 2 | 59 |
|----------------------------------|----|
| 8.2.5.4. PFS vs HEMOGLOBIN | 60 |
| 8.2.5.5. PFS vs LIVER METASTASIS | 61 |
| 8.2.6. OS | 62 |
| 8.2.6.1. OS vs Age>70 | 64 |
| 8.2.6.2. OS vs Renal Impairment | 64 |
| 8.2.6.3. OS vs ECOG 2 | 66 |
| 8.2.6.4. OS vs HEMOGLOBIN | 67 |
| 8.2.6.5. OS vs LIVER METASTASIS | 68 |
| 9. Safety analysis | 69 |
| 9.1. Annex 1 | 74 |

The database was locked down on XXX.

#### 2. STUDY DESIGN

The SOGUG-AUREA study is a multicenter, open labelled, single arm, Phase II clinical trial of atezolizumab in combination of split-dose cisplatin plus gemcitabine in patients with locally advanced or metastatic urothelial carcinoma (additional details on the eligibility criteria of the study are found in section 6 of the study protocol).

The design includes screening phase, combined treatment initial phase, monotherapy treatment phase, follow-up phase and translational research with biopsies, blood samples and faecal samples.

The dose scheme includes the initial dose of atezolizumab (1200 mg) intravenously administered every 21 days (one cycle) up to disease progression, unacceptable toxicity or absence of clinical benefit. Dose adjustment or dose reductions of atezolizumab are not expected. Additional information on the treatment, modifications, and dose delays is available in section 7 of the study protocol. SOGUG-AUREA is an Investigator Initiated Study, the Sponsor will supply Atezolizumab for up to 24 months of treatment for each patient. For those patients in which the PI considers that the best option for the patient is continuing atezolizumab for more than 24 months, available commercial Site supplies should be used, after managed local administrative regulation.

# 3. SCREENING FAILURE

Table 1: Frequency screening failures

| Overall | Overall (N=) |
|---------------------------|--------------|
| Screening Failing | |
| No | |
| Yes | |
| Screening Failure Specify | |

Table 2: List of patients with screening failure

| Patient number | Screening Failing | Screening Failure Specify |
|----------------|-------------------|---------------------------|

Table 3: Patients without screening failure by hospital

| Overall | Overall (N=) |
|------------------------------------------------|--------------|
| Hospital | |
| COMPLEJO HOSPITALARIO DE JAÉN | |
| COMPLEXO HOSPITALARIO UNIVERSITARIO DE OURENSE | |
| CONSORCIO HOSPITALARIO PROVINCIAL DE CASTELLÓN | |
| HOSPITAL CLÍNICO SAN CARLOS | |
| HOSPITAL DE LA SANTA CREU I SANT PAU | |
| HOSPITAL SON LLATZER | |
| HOSPITAL UNIVERSITARIO 12 DE OCTUBRE | |
| HOSPITAL UNIVERSITARIO CENTRAL DE ASTURIAS | |
| HOSPITAL UNIVERSITARIO INSULAR DE GRAN CANARIA | |
| HOSPITAL UNIVERSITARIO LA PAZ | |
| HOSPITAL VIRGEN DE LA SALUD | |
| INSTITUT CATALÀ D'ONCOLOGIA L'HOSPITALET ICO | |

## 4. STUDY POPULATIONS

#### 4.1. INTENT-TO-TREAT

Intent-To-Treat (ITT): All patients that have been enrolled in the trial.

Table 4: ITT population

| Overall | Overall (N=) |
|----------------------------|--------------|
| Intent-to-treat population | |
| No | |
| Yes | |
| ITT population exclusion | |
| reason | |
| NA | |
| Screening Failure | |

Table 5: ITT exclusion reason

| Patient number | Intent-to-treat population | ITT population exclusion reason |
|---|---|---|

### 4.2. PER PROTOCOL

Evaluable population **per protocol (PP)**: All patients fulfilling all eligibility criteria without any protocol deviation that makes the patient invalid for the primary endpoint evaluation.

Table 6: PP population

| Overall | Overall (N=) |
|-------------------------|--------------|
| Per protocol population | |
| No | |
| Yes | |
| PP population exclusion | |
| reason | |
| NA | |
| Screening Failure | |

Table 7: PP exclusion reason

| Patient number | Per protocol population | PP population exclusion reason |
|----------------|-------------------------|--------------------------------|

## 4.3. SAFETY POPULATION

**Safety population (SP)**: All patients receiving at least one dose of the study treatments.

Table 8: Safety population

| Overall | Overall (N=) |
|-----------------------------|--------------|
| Safety population | |
| No | _ |
| Yes | |
| Safety population exclusion | _ |
| reason | |
| NA | |
| Screening Failure | |

Table 9: Safety exclusion reason

| Patient number | Safety population | Safety population exclusion reason |
|----------------|-------------------|------------------------------------|

## 5. BASAL INFORMATION

This section is carried out in the ITT population (N = XX patients).

#### **5.1.** Non-cisplatin eligible

Table 10: Frequency non-cisplatin eligible

| Overall | Overall (N=) |
|------------------------------------------------|--------------|
| ECOG 2 | |
| Yes | |
| No | |
| Age > 70 years | |
| Yes | |
| No | |
| Creatinine clearance >30 µmol/L and <60 µmol/L | |
| Yes | |
| No | |
| Other non-cisplatino elegible reason | |
| Yes | |
| No | |
| Specify other non-cisplatino elegible reason | |

Table 11: Frequency non-cisplatin eligible combined

| Overall | Overall (N=) |
|------------------------------------------|--------------|
| Non-cisplatino elegible reasons combined | |

# **5.2.** CANCER HISTORY 5.2.1. PRIMARY CANCER

Table 12: Frequency primary cancer location

| Overall | Overall (N=) |
|--------------|--------------|
| Cancer | |
| Location | |
| Urothelial | |
| cancer | |
| Location | |
| Specify | |
| Renal pelvis | |
| Ureter | |
| Bladder | |
| Urethra | |

Table 13: Frequency TNM status at diagnosis

| Overall | Overall (N=) |
|-----------------|--------------|
| Initial T Stage | |
| T1 | |
| T2 | |
| T2a | |
| T2b | |
| T3 | |
| T3b | |
| T4 | |
| T4a | |
| T4b | |
| Tis | |
| Ta | |
| Tx | |
| Initial N Stage | |
| N0 | |
| N1 | |
| N2 | |
| N3 | |
| Nx | |
| Initial M Stage | |
| M0 | |
| M1 | |
| М1а | |
| M1b | |
| Mx | |
| Cancer Stage | |
| 0a | |
| 0is | |
| 1 | |
| <u> </u> | |
| III | |

| Overall | Overall (N=) |
|-----------------------|--------------|
| IIIA | |
| IIIB | |
| IV | |
| IVA | |
| IVB | |
| Unknown | |
| Differentiation | |
| Well differentiated | |
| Moderately | |
| differentiated | |
| Poorly differentiated | |
| Undifferentiated | |
| Unknown | |
| Cancer History Grade | |
| High | |
| Low | <u> </u> |
| Unknown | |

Table 14: List of patients with Unknown Cancer Stage

| Patient Number | Hospital | Cancer Stage |
|----------------|-------------------------------|--------------|
| 004-007 | HOSPITAL UNIVERSITARIO LA PAZ | Unknown |

Table 15: Frequency metastasis location

| | Overall |
|-------------------------|-------------------|
| Overall | Overall<br>(N=66) |
| Metastasis | (14-00) |
| Yes | 28 (42.4%) |
| No | 38 (57.6%) |
| Metastasis Liver | 00 (01:070) |
| NA | 61 (92.4%) |
| Liver | 5 (7.6%) |
| Metastasis Peritoneum | |
| NA | 64 (97.0%) |
| Peritoneum | 2 (3.0%) |
| Metastasis Pleura | _ (0:0::) |
| NA | 65 (98.5%) |
| Pleura | 1 (1.5%) |
| Metastasis Lung | . ( ) |
| NA | 52 (78.8%) |
| Lung | 14 (21.2%) |
| Metastasis Kidney | (= ::= :: / |
| NA | 65 (98.5%) |
| Kidney | 1 (1.5%) |
| Metastasis Bone | , , |
| NA | 60 (90.9%) |
| Bone | 6 (9.1%) |
| Metastasis Renal | , |
| NA | 65 (98.5%) |
| Renal | 1 (1.5%) |
| Metastasis Soft tissues | , |
| NA | 65 (98.5%) |
| Soft tissues | 1 (1.5%) |
| Metastasis Skin | |
| NA | 65 (98.5%) |
| Skin | 1 (1.5%) |
| Metastasis Lymph | |
| nodes | |
| NA | 48 (72.7%) |
| Lymph nodes | 18 (27.3%) |
| Metastasis Other | |
| NA | 64 (97.0%) |
| Other | 2 (3.0%) |
| Metastasis Other | |
| specify | 0.4 (0= 00() |
| NA | 64 (97.0%) |
| Adrenal | 1 (1.5%) |
| Suprarrenal | 1 (1.5%) |

Table 16: Frequency current metastasis location

| | 0 " (1) |
|---------------------------------|--------------|
| Overall | Overall (N=) |
| Current status | |
| Locally advanced | |
| Metastasic | |
| Current Metastasis Colon | |
| NA | |
| Colon | |
| Current Metastasis Pleural | |
| effusion | |
| NA | |
| Pleural effusion | |
| Current Metastasis Liver | |
| NA | |
| Liver | |
| Current Metastasis Large | |
| intestine | |
| NA | |
| Large intestine | |
| Current Metastasis Mediastinum | |
| NA | |
| Mediastinum | |
| Current Metastasis Pancreas | |
| NA | |
| Pancreas | |
| Current Metastasis Peritoneum | |
| NA | |
| Peritoneum | |
| Current Metastasis Lung | |
| NA | |
| Lung | |
| Current Metastasis Kidney | |
| NA | |
| Kidney | |
| Current Metastasis Bone | |
| NA | |
| Bone | |
| Current Metastasis Renal | |
| NA | |
| Renal | |
| Current Metastasis Soft tissues | |
| NA | |
| Soft tissues | |
| Current Metastasis Skin | |
| NA<br>NA | |
| Skin | |
| Current Metastasis Jejunum | |
| NA | |
| Jejunum | |
| Current Metastasis Lymph nodes | |
| NA | |
| Lymph nodes | |

| Overall | Overall (N=) |
|-----------------------------------------|--------------|
| <b>Current Metastasis Other</b> | |
| NA | |
| Other | |
| <b>Current Metastasis Other specify</b> | |
| NA | |
| Adrenal | |
| Paraaortic | |
| Vagina | |

Table 17: Frequency calculated metastasis location

| Overall | Overall<br>(N=) |
|---------------------------------------------|-----------------|
| Lung - Metastasis | • |
| No | |
| Yes | |
| Other - Adrenal - Metastasis | |
| No | |
| Yes | |
| Renal - Metastasis | |
| No | |
| Yes | |
| Peritoneum - Metastasis | |
| No | |
| Yes | |
| Lymph nodes - Metastasis | |
| No | |
| Yes | |
| Mediastinum - Metastasis | |
| No | |
| Yes | |
| Diaphragma - Metastasis | |
| No | |
| Yes | |
| Other - left cardiophrenic fat - Metastasis | |
| No | |
| Yes | |
| Liver - Metastasis | |
| No | |
| Yes | |
| Kidney - Metastasis | |
| No | |
| Yes | |
| Bone - Metastasis | |
| No | |
| Yes | |
| Other Metastasis | |
| No | |
| Yes | |
| Large intestine - Metastasis | |

| Overall | Overall<br>(N=) |
|--------------------------------------|-----------------|
| No | (* * / |
| Yes | |
| Jejunum - Metastasis | |
| No | |
| Yes | |
| Mesenterium - Metastasis | |
| No | |
| Yes | |
| Other - penile implant - Metastasis | |
| No | |
| Yes | |
| Ileus - Metastasis | |
| No | |
| Yes | |
| Other - supraclavicular - Metastasis | |
| No | |
| Yes | |
| Other-inter-aortocava - Metastasis | |
| No | |
| Yes | |
| Pleural effusion - Metastasis | |
| No | |
| Yes | |
| Pleura - Metastasis | |
| No | |
| Yes | |
| Pancreas - Metastasis | |
| No | |
| Yes Other - Gallbladder - Metastasis | |
| No | |
| Yes | |
| Other: omentum - Metastasis | |
| No | |
| Yes | |
| Soft tissues - Metastasis | |
| No | |
| Yes | |
| Ascites - Metastasis | |
| No | |
| Yes | |
| Skin - Metastasis | |
| No | |
| Yes | |
| Colon - Metastasis | |
| No | |
| Yes | |
| 100 | |

Table 18: Frequency treatments

| Overall | Overall (N=) |
|------------------------------|--------------|
| Surgery | |
| Yes | |
| No | |
| Primary Surgery | |
| NA | |
| Yes | |
| Surgery Outcome | |
| NA | |
| R0 | |
| R1 | |
| R2 | |
| Unknown | |
| Radiotherapy | |
| Yes | |
| No | |
| Radiotherapy cycles | |
| NA | |
| 1 | |
| 2 | |
| Unknown | |
| Radiotherapy cycles | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Radiotherapy Cumulative dose | |
| (Gy) | |
| Radiotherapy Cumulative dose | |
| (Gy) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range Previous treatment | |
| Yes | |
| No | |
| Unknown | |
| Other cancer history | |
| Yes | |
| No | |
| Cancer History Type | |
| Cancer History Treatment | |
| | 5 40 5 == |

| Overall | Overall (N=) |
|---------|--------------|

## 5.3. DEMOGRAPHIC DATA

Table 19: Frequency demographic data

| 0 | O |
|---------------------------------|--------------|
| Overall | Overall (N=) |
| Patient Age N | |
| Mean (95%CI) SD | |
| Median (95%CI) | |
| Range<br>Gender | |
| Male | |
| Female | |
| Weight (Kg) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Race | |
| Caucasian | |
| Latin | |
| Systolic Blood Pressure (mmHG) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Diastolic Blood Pressure (mmHG) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Temperature (°C) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Height (cm) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Respiratory rate (breaths per | |
| minute) | |
| N | |
| Mean (95%CI) | |
| SD | |

| Overall | Overall (N=) |
|-------------------------|--------------|
| Median (95%CI) | |
| Range | |
| Pulse rate (bpm) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Body Mass Index (kg/m2) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| ECOG | |
| 0 | |
| 1 | |
| 2 | |
| Physical exam | |
| Normal | |
| Abnormal | |

## 5.4. COMORBIDITIES AND CONCOMITANT MEDICATION

Table 20: Frequency comorbidities and concomitant medication

| Overall | Overall (N=) |
|---------------|--------------|
| Comorbidities | |
| No | |
| Yes | |
| Concomitant | |
| Medication | |
| No | |
| Yes | |

Table 21: Frequency comorbidities in patients

| Comorbidities | N | % |
|---------------|---|---|

\*Some patients can have several comorbidities

Table 22: Frequency other comorbidities in patients

| Comorbidities | N | % |
|---------------|---|---|

\*Some patients can have several comorbidities

Table 23: Frequency concomitant medication in patients

| Concomitant medication | N | % |
|------------------------|---|---|

<sup>\*</sup>Some patients can have several concomitant medications

Table 24: Frequency other concomitant medication in patients

| Other concomitant medication | N | % |
|------------------------------|---|---|

<sup>\*</sup>Some patients can have several concomitant medications

#### 5.5. HEMATOLOGY AND COAGULATION

Table 25: Frequency hematology and coagulation

| Overall | Overall (N=) |
|---------------------------|--------------|
| Hemoglobin Value (g/dL) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Platelets Value (10e3/µL) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Neutrophils Value | |
| (10e3/µL) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |

## 5.6. BIOCHEMISTRY, SEROLOGY AND THYROID FUNCTION

Table 26: Frequency biochemistry, serology and thyroid function

| - " | - " " " " |
|-----------------------------|--------------|
| Overall | Overall (N=) |
| Creatinine Value (mg/dL) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Creatinine Clearing Value | |
| (ml/min) | |
| N (050( OL) | |
| Mean (95%CI) | |
| SD (050/ O)) | |
| Median (95%CI) | |
| Range | |
| Bilirubin Value (mg/dL) | |
| N<br>Macro (05% CI) | |
| Mean (95%CI) | |
| SD<br>Modion (05% CI) | |
| Median (95%CI) | |
| Range Bilirubin Value < ULN | |
| Yes | |
| ALT Value (U/L) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| ALT Value < ULN | |
| No | |
| Yes | |
| AST Value (U/L) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| AST Value < ULN | |
| No | |
| Yes | |
| GGT Value (U/L) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| GGT Value < ULN | |
| No | |

| Overall | Overall (N=) |
|---------|--------------|
| Yes | |
| Unknown | |

## **5.7.** OTHER DETERMINATIONS

Table 27: Frequency other determinations

| Overall | Overall (N=) |
|----------------------|--------------|
| Urine Analysis ND | |
| Done | |
| Not done | |
| Urine Analysis | |
| Missing data | |
| Negative | |
| Traces | |
| +1 | |
| +2 | |
| +3 | |
| +4 | |
| Urine Analysis Blood | |
| NA | |
| Positive | |
| Negative | |
| Urine Analysis | |
| Glucose | |
| NA | |
| Normal | |
| Abnormal | |
| Urine Analysis | |
| Protein | |
| NA | |
| Positive | |
| Negative | |
| Pregnancy Test Value | |
| NA | |
| Negative | |
| Unknown | |
| Electrocardiogram | |
| Done | |
| Ecg Value | |
| Normal | |
| Abnormal | |
| FEVI | |
| Done | |
| Not done | |
| FEVI Value | |
| NA | |
| Normal | |
| Abnormal | |

#### 6. TREATMENT COMPLIANCE

The following analyses in this section are carried out in the safety population (N = XX patients).

# 6.1. INITIAL PHASE: COMBINED TREATMENT (C1-C6) ATEZOLIZUMAB, CISPLATIN AND GEMCITABINE

Table 28: Adherence to atezolizumab, cisplatin and gemcitabine

| Overall | Overall (N=) |
|--------------------------------------------------------------|--------------|
| Number of cycles administered (Initial phase) - Atezolizumab | Overam (iv ) |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Number of cycles administered (Initial phase) - Atezolizumab | |
| 1 | |
| 2 | |
| 3 | |
| 4 | |
| 5 | |
| 6 | |
| Atezolizumab treatment duration (months) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Number of cycles administered (partial/complete) - Cisplatin | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Number of cycles administered (complete) - Cisplatin | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Number of cycles administered (partial/complete) - Cisplatin | |
| 1 | |
| 2 | |
| 3 | |
| 4 | |
| 5 | |
| 6 | |
| Number of cycles administered (complete) - Cisplatin | |
| 0 | |

| Q II | O |
|---|---|
| Overall | Overall (N=) |
| 1 | |
| 2 | |
| 3 | |
| 4 | |
| 5 | |
| 6 | |
| Cisplatin treatment duration (months) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Number of cycles administered (partial/complete) - Gemcitabine | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Number of cycles administered (complete) - Gemcitabine | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Number of cycles administered (partial/complete) - Gemcitabine | |
| 2 | |
| 3 | |
| 4 | |
| 5 | |
| 6 | |
| Number of cycles administered (complete) - Gemcitabine | |
| 0 | |
| _ 1 | |
| 2 | |
| 3 | |
| 4 | |
| 5 | |
| 6 | |
| Gemcitabine treatment duration (months) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |

Table 29: Atezolizumab, cisplatin and gemcitabine omissions

| | O 11 /h1 ) |
|---|---|
| Overall Advantage of the Control of | Overall (N=) |
| Omission (Initial phase) - Atezolizumab | |
| No | |
| Yes | |
| Number of patients with omission (Initial phase) - Atezolizumab | |
| N (STOCK OF ) | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Number of patients with omissions (Initial phase) - Atezolizumab | |
| 0 | |
| Omission - Cisplatin | |
| No | |
| Yes | |
| Number of patients with an omission - Cisplatin | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Number of patients with two omissions - Cisplatin | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Number of patients with an omission - Cisplatin | |
| 0 | |
| 1 | |
| 2 | |
| 3 | |
| 5 | |
| Number of patients with two omissions - Cisplatin | |
| 0 | |
| 1 | |
| Omission - Gemcitabine | |
| No | |
| Yes | |
| Number of patients with an omission - Gemcitabine | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Number of patients with two omissions - Gemcitabine | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |

| Overall | Overall (N=) |
|-----------------------------------------------------|--------------|
| Range | |
| Number of patients with an omission - Gemcitabine | |
| 0 | |
| 1 | |
| 2 | |
| 3 | |
| 5 | |
| Number of patients with two omissions - Gemcitabine | |
| 0 | |
| 1 | _ |

Table 30: List of omissions reasons

| Atezolizumab - Omission reason | | N | % |
|--------------------------------|---|---|---|
| Other | | | |
| Cisplatin - Omission reason | N | | % |
| AE | | | |
| Other | | | |
| Gemcitabine - Omission reaso | n | N | % |
| AE | | | |
| Other | | | |

Table 31: List of other omissions reasons specify

| Atezolizumab - Omission reason | | | % |
|--------------------------------|---|---|--------|
| Cisplatin - Omission reason N | | % | |
| Gemcitabine - Omission reason | N | % | ,<br>D |

Table 32: Atezolizumab, cisplatin and gemcitabine delays

| Overall | Overall (N=) |
|---|---|
| Delay (Initial phase) - Atezolizumab | <b>O</b> 1010 (11 ) |
| No | |
| Yes | |
| Number of cycles with delay (Initial phase) - Atezolizumab | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Number of cycles with delay (Initial phase) - Atezolizumab | |
| 0 | |
| 2 | |
| 1 | |
| 3 | |
| 4 | |
| Delay | |
| No | |
| Yes | |
| Number of cycles with a delay - Cisplatin | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Number of cycles with two delays - Cisplatin | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Number of cycles with a delay - Cisplatin | |
| 0 | |
| 1 | |
| 2 | |
| 3 | |
| 4 | |
| Number of cycles with two delays - Cisplatin | |
| 0 | |
| 1 | |
| 2 | |
| Delay - Gemcitabine | |
| No | |
| Yes | |
| Number of cycles with a delay - Gemcitabine | |
| N | |
| Mean (95%CI) | |
| SD<br>Madian (05% CI) | |
| Median (95%CI) | |
| Range | |
| Number of cycles with two delays - Gemcitabine | |

| Overall | Overall (N=) |
|------------------------------------------------|--------------|
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Number of cycles with a delay - Gemcitabine | |
| 0 | |
| 1 | |
| 2 | |
| 3 | |
| 4 | |
| Number of cycles with two delays - Gemcitabine | |
| 0 | |
| 1 | |
| 2 | |

Table 33: List of delay reasons

| Atezolizumab - Delay reaso | on | N | 9, | 6 |
|----------------------------|----|---|----|---|
| AE | | | | |
| Other | | | | |
| Cisplatin - Delay reason | N | | % | |
| AE | | | | |
| Other | | | | |
| Gemcitabine - Delay reaso | n | N | % | |
| AE | | | | |
| Other | | | | |

Table 34: List of other delay reasons

| Atezolizumab - Delay reason | N | % |
|-----------------------------|---|---|
| Cisplatin - Delay reason | N | % |
| Gemcitabine - Delay reason | N | % |

Table 35: Cisplatin and gemcitabine dose decrease

| Overall | Overall (N=) |
|----------------------------------------------------|--------------|
| Dose reduction | |
| No | |
| Yes | |
| Number of cycles with a dose reduction - Cisplatin | |
| N | |

| Overall | Overall (N=) |
|---------------------------------------------------------|--------------|
| Mean (95%CI) | 0 101u (11 ) |
| SD | |
| Median (95%CI) | |
| Range | |
| Number of cycles with two dose reductions - Cisplatin | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Number of cycles with a dose reduction - Cisplatin | |
| 0 | |
| 1 | |
| 2 | |
| Number of cycles with two dose reductions - Cisplatin | |
| 0 | |
| Minimum dose in dose reductions - Cisplatin | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Dose reduction - Gemcitabine | |
| No | |
| Yes | |
| Number of cycles with a dose reduction - Gemcitabine | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Number of cycles with two dose reductions - Gemcitabine | |
| <u>N</u> | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Number of cycles with a dose reduction - Gemcitabine | |
| 0 | |
| 1 | |
| 2 | |
| Number of cycles with two dose reductions - Gemcitabine | |
| 0 | |
| Minimum dose in dose reductions - Gemcitabine | |
| N (270(2)) | |
| Mean (95%CI) | |
| SD (CTO) | |
| Median (95%CI) | |
| Range | |

Table 36: List of dose decrease reasons

| Cisplatin - Dose reduction reason | N | % |
|-------------------------------------|---|---|
| AE | | |
| Gemcitabine - Dose reduction reason | N | % |
| AE | | |
| Other | | |

Table 37: List of other dose decrease reasons (AEs)

| Cisplatin - Dose reduction reason | N | % |
|-------------------------------------|---|---|
| Gemcitabine - Dose reduction reason | N | % |

Table 38: Cisplatin and gemcitabine re-scalation after dose reduction

| Overall | Overall (N=) |
|---|---|
| Dose re-scalation after dose reduction | |
| No | |
| Yes | |
| Number of cycles with a re-scalation after dose reduction - Cisplatin | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Number of cycles with two re-scalation after dose reduction - Cisplatin | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Number of cycles with a re-scalation after dose reduction - Cisplatin | |
| 0 | |
| 1 | |
| Number of cycles with two re-scalation after dose reduction - Cisplatin | |
| 0 | |
| Minimum dose in dose re-scalation after dose reduction - Cisplatin | |
| N . | |
| Mean | |
| SD | |
| Median | |
| Range | |
| Dose re-scalation after dose reduction - Gemcitabine | |
| No | |
| Yes | |
| Number of cycles with a re-scalation after dose reduction - Gemcitabine | |

| Overall | Overall (N=) |
|---|---|
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Number of cycles with two re-scalation after dose reduction - | |
| Gemcitabine | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Number of cycles with a re-scalation after dose reduction - Gemcitabine | |
| 0 | |
| Number of cycles with two re-scalation after dose reduction - | |
| Gemcitabine | |
| 0 | |
| Minimum dose in dose re-scalation after dose reduction - Gemcitabine | |
| N . | |
| Mean | |
| SD | |
| Median | |
| Range | |

Table 39: List of re-scalation after dose reduction reasons

| Cisplatin - Re-scalation after dose reduction reason | N | % |
|--------------------------------------------------------|---|---|
| Gemcitabine - Re-scalation after dose reduction reason | N | % |

# **6.2.** Monotherapy phase: Adherence to atezolizumab and entire treatment

Table 40: Adherence to atezolizumab, monotherapy phase and entire treatment

| Number of cycles administered (Monotherapy phase) - Atezolizumab N Mean (95%CI) SD Median (95%CI) Range Number of cycles administered (Monotherapy phase) - Atezolizumab 0 1 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab N Mean (95%CI) SD Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab 1 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab 1 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) | Overall | Overall (N=) |
|---|---|---|
| New Median (95%CI) SD Median (95%CI) Range Number of cycles administered (Monotherapy phase) - Atezolizumab 0 1 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab N Mean (95%CI) SD Median (95%CI) SD Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab 1 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab 1 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) SD Median (95%CI) | | Overall (N=) |
| Mean (95%CI) SD Median (95%CI) Range Number of cycles administered (Monotherapy phase) - Atezolizumab 0 1 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab N Mean (95%CI) SD Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab 1 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) SD Median (95%CI) SD Median (95%CI) SD Median (95%CI) | | |
| SD Median (95%CI) Range Number of cycles administered (Monotherapy phase) - Atezolizumab 0 1 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab N Mean (95%CI) SD Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab 1 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) SD Median (95%CI) SD Median (95%CI) | | |
| Median (95%CI) Range Number of cycles administered (Monotherapy phase) - Atezolizumab 0 1 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab N Mean (95%CI) SD Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab 1 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab 1 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) SD Median (95%CI) | | |
| Range Number of cycles administered (Monotherapy phase) - Atezolizumab 0 1 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab N Mean (95%CI) SD Median (95%CI) SD Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab 1 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) SD Median (95%CI) SD Median (95%CI) SD Median (95%CI) | | |
| Number of cycles administered (Monotherapy phase) - Atezolizumab 0 1 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab N Mean (95%CI) SD Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab 1 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) SD Median (95%CI) SD Median (95%CI) | | |
| 0 1 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab N Mean (95%CI) SD Median (95%CI) SD Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab 1 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) SD Median (95%CI) SD | | |
| 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab N Mean (95%CI) SD Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab 1 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) SD Median (95%CI) SD Median (95%CI) | | |
| Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab N Mean (95%CI) SD Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab 1 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) SD Median (95%CI) | 1 | |
| Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab N Mean (95%CI) SD Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab 1 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) SD Median (95%CI) SD Median (95%CI) | 2 | |
| N Mean (95%CI) SD Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab N Mean (95%CI) SD Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab 1 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) SD Median (95%CI) | 3 | |
| N Mean (95%CI) SD Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab N Mean (95%CI) SD Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab 1 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) SD Median (95%CI) | | |
| Mean (95%CI) SD Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab N Mean (95%CI) SD Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab 1 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) SD Median (95%CI) | Atezolizumab treatment duration (months) | |
| Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab N Mean (95%CI) SD Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab 1 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) SD Median (95%CI) | N | |
| Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab N Mean (95%CI) SD Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab 1 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) | | |
| Number of cycles administered (Entire treatment) - Atezolizumab N Mean (95%CI) SD Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab 1 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) | | |
| Number of cycles administered (Entire treatment) - Atezolizumab N Mean (95%CI) SD Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab 1 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) | Median (95%CI) | |
| N Mean (95%CI) SD Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab 1 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) | | |
| Mean (95%CI) SD Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab 1 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) | | |
| SD Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab 1 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) | | |
| Median (95%CI) Range Number of cycles administered (Entire treatment) - Atezolizumab 1 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) | | |
| Range Number of cycles administered (Entire treatment) - Atezolizumab 1 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) | | |
| Number of cycles administered (Entire treatment) - Atezolizumab 1 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) | | |
| 1 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) | | |
| 2 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) | - | |
| 3 Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) | | |
| Atezolizumab treatment duration (months) N Mean (95%CI) SD Median (95%CI) | | |
| N<br>Mean (95%CI)<br>SD<br>Median (95%CI) | | |
| N<br>Mean (95%CI)<br>SD<br>Median (95%CI) | Atezolizumah treatment duration (months) | |
| SD<br>Median (95%CI) | | |
| SD<br>Median (95%CI) | Mean (95%CI) | |
| Median (95%CI) | | |
| | Range | |
Table 41: Atezolizumab omissions, monotherapy phase and entire treatment

| Overall | Overall (N=) |
|---|---|
| Omission (Monotherapy phase) - Atezolizumab | <b>5</b> * 5 * 5 * 5 * 7 |
| No | |
| Yes | |
| Number of cycles with omission (Monotherapy phase) - Atezolizumab | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Number of cycles with omissions (Monotherapy phase) - Atezolizumab | |
| 0 | |
| Omission (Entire treatment) - Atezolizumab | |
| No | |
| Yes | |
| Number of cycles with omission (Entire treatment) - Atezolizumab | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Number of cycles with omissions (Entire treatment) - Atezolizumab | |
| 0 | |

Table 42: List of omissions reasons

| Atezolizumab - Omission reason (Monotherapy) | N | % |
|---------------------------------------------------|---|---|
| Atezolizumab - Omission reason (Entire treatment) | N | % |
| , | | |

Table 43: List of omissions reasons specify

| Atezolizumab - Omission reason (Entire treatment) | N | % |
|---------------------------------------------------|---|---|

Table 44: Atezolizumab delays, monotherapy phase and entire treatment

| Overall | Overall (N=) |
|---|---|
| Delay (Monotherapy phase) - Atezolizumab | , , |
| No | |
| Yes | |
| Number of cycles with delay (Monotherapy phase) - Atezolizumab | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Number of cycles with delay (Monotherapy phase) - Atezolizumab | |
| 0 | |
| 2 | |
| Delay (Entire treatment) - Atezolizumab | |
| No | |
| Yes | |
| Number of cycles with delay (Entire treatment) - Atezolizumab | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |
| Number of cycles with delay (Entire treatment) - Atezolizumab | |
| 0 | |
| 1 | |
| 2 | |

Table 45: List of delay reasons

| Atezolizumab - Delay reason (Monotherapy) | N | % |
|------------------------------------------------|---|---|
| Atezolizumab - Delay reason (Entire treatment) | N | % |

Table 46: List of other delay reasons

| Atezolizumab - Delay reason (Monotherapy) | N | % |
|------------------------------------------------|---|---|
| Atezolizumab - Delay reason (Entire Treatment) | N | % |

## 7. END OF TREATMENT

The following analyses in this section are carried out in the safety population (N = XX patients).

Table 47: End of treatment

| Overall | Overall (N=) |
|----------------------------------------------|--------------|
| End of Atezolizumab Treatment Reason | |
| Progression according RECIST 1.1 | |
| Death | |
| Study treatment completion | |
| AE not related to the treatment study | |
| Unnacceptable toxicity | |
| Investigator decision | |
| Withdraw consent | |
| Other | |
| End of Atezolizumab Treatment Reason Specify | |
| End of Cisplatin Treatment Reason | |
| Study treatment completion | |
| Unnacceptable toxicity | |
| Progression according RECIST 1.1 | |
| Death | |
| AE not related to the treatment study | |
| Investigator decision | |
| Withdraw consent | |
| Other | |
| End of Gemcitabine Treatment Reason | |
| Study treatment completion | |
| Unnacceptable toxicity | |
| Progression according RECIST 1.1 | |
| Death | |
| AE not related to the treatment study | |
| Investigator decision | |
| Withdraw consent | |
| Other | |

Note: the following reasons have been recoded to minimize categories - Kidney function impairment/Urinary tract infection/: AE not related to the treatment study

Table 48: End of treatment (Grouped to minimize categories)

| Treatment | Atezolizumab<br>(N=) | Cisplatin<br>(N=) | Gemcitabine<br>(N=) | Total (N=) |
|---|---|---|---|---|
| End of treatment reason | | | | |
| Study treatment | | | | _ |
| completion | | | | |
| Progression disease | | | | |
| Unnacceptable toxicity | | | | |

| Treatment | Atezolizumab<br>(N=) | Cisplatin<br>(N=) | Gemcitabine<br>(N=) | Total (N=) |
|---|---|---|---|---|
| Death | | | | |
| AE not related to the | | | | |
| treatment study | | | | |
| Investigator decision | | | | |
| Withdraw consent | · | · | _ | · |
| Other | | | | |

 $^{\it Note}$ : the following reasons have been recoded to minimize categories - Symptomatic deterioration/Progression according RECIST 1.1/Clinical Progression: Progression disease

Figure 1: Atezolizumab treatment discontinuation

Figure 2: Cisplatin treatment discontinuation

Figure 3: Gemcitabine treatment discontinuation

# 8. Efficacy analysis

The following analyses in this section are carried out in the Per Protocol population (N = XX patients).

### 8.1. PRIMARY OBJECTIVE

### 8.1.1. Overall response rate (ORR)

To evaluate the preliminary efficacy of atezolizumab plus split-dose gemcitabine and cisplatin (GC) for the first-line setting, in patients with histologically confirmed advanced (locally advanced and metastatic) urothelial cancer in terms of overall response rate (ORR) assessed by the investigator using the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

**Overall Response Rate (ORR)**: Assessed by the investigator using the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. This will be considered as the percentage/proportion of patients with confirmed complete response (CR) or partial response (PR) as their overall best response throughout the study period.

Table 49: Frequency best overall response

| Best OR Confirmed | N | % | 95%CI |
|-------------------|---|---|-------|
| CR | | | |
| PR | | | |
| SD | | | |
| PD | | | |
| NE/UK | | | |
| UK | | | |
| Total | | | |

Table 50: List of patients with NE/UK as best overall response

| Patient number | Best OR<br>Confirmed | Resp. 1.1 | Tumor<br>Assessment<br>Target Sum | Status | EOS Date | End of Trial<br>Reason | Exitus Reason | Exitus Reason<br>Specify |
|---|---|---|---|---|---|---|---|---|

Table 51: Frequency best overall response without UK/NE

| Best OR Confirmed | N | % | 95%CI |
|-------------------|--------|----------|-------|
| CR | | | |
| | Page 4 | 15 of 77 | |

| Best OR Confirmed | N | % | 95%CI |
|-------------------|---|---|-------|
| PR | | | |
| SD | | | |
| PD | | | |
| NE | | | |
| UK | | | |
| Total | | | |

Table 52: List of patients with CR/PR as best overall response

| Patient number | Hospital | Best OR Confirmed |
|----------------|----------|-------------------|

Table 53: Frequency overall response rate

| Overall Response Rate (confirmed) | N | % | 95%CI |
|-----------------------------------|---|---|-------|
| Yes (CR/PR) | | | |
| No | | | |
| Total | | | |

Table 54: Frequency overall response rate without UK/NE

| Overall Response Rate (confirmed) | N | % | 95%CI |
|-----------------------------------|---|---|-------|
| Yes (CR/PR) | | | |
| No | | | |
| Total | | | |

Figure 4: Waterfall plot

#### 8.1.1.1. ORR vs Age>70

Table 1: Age>70 by Overall response rate

| Age > 70 years | No (N=) | Yes (N=) | Total (N=) | p-value |
|---|---|---|---|---|
| Overall Response Rate (confirmed) | | | | |
| N | | | | |
| No | | | | |
| Yes (CR/PR) | | | | |

### (1) Fisher's exact test

(\*) The percentages take into account missing data, the p-values do not

Table 2: Age>70 by Overall response rate without UK/NE

| Age > 70 years | No (N=) | Yes (N=) | Total (N=) | p-value |
|---|---|---|---|---|
| Overall Response Rate (confirmed) | | | | |
| N | | | | |
| Yes (CR/PR) | | | | |
| No | | | | |

### (1) Fisher's exact test

#### 8.1.1.2. ORR VS RENAL IMPAIRMENT

Table 3: Renal Impairment by Overall response rate

| Creatinine clearance >30 µmol/L and <60 µmol/L | No (N=) | Yes (N=) | Total (N=) | p-value |
|---|---|---|---|---|
| Overall Response Rate (confirmed) | | | | |
| N | | | | |
| No | | | | |
| Yes (CR/PR) | | | | |

### (1) Fisher's exact test

(\*) The percentages take into account missing data, the p-values do not

Table 4: Renal Impairment by Overall response rate without UK/NE

| Creatinine clearance >30 µmol/L and <60 µmol/L | No (N=) | Yes (N=) | Total (N=) | p-value |
|---|---|---|---|---|
| Overall Response Rate (confirmed) | | | | |
| N | | | | |
| Yes (CR/PR) | | | | |
| No | | | | |

### (1) Fisher's exact test

#### 8.1.1.3. ORR vs ECOG 2

Table 5: ECOG 2 by Overall response rate

| ECOG 2 | No (N=) | Yes (N=) | Total (N=) | p-value |
|---|---|---|---|---|
| Overall Response Rate (confirmed | l) | | | |
| N | 51 | 15 | 66 | |
| No | 26 (51.0%) | 8 (53.3%) | 34 (51.5%) | |
| Yes (CR/PR) | 25 (49.0%) | 7 (46.7%) | 32 (48.5%) | |

<sup>(1)</sup> Fisher's exact test

(\*) The percentages take into account missing data, the p-values do not

Table 6: ECOG 2 by Overall response rate without UK/NE

| ECOG 2 | No (N=) | Yes (N=) | Total (N=) | p-value |
|---|---|---|---|---|
| Overall Response Rate (confirmed) | | | | |
| N | | | | |
| Yes (CR/PR) | | | | |
| No | | | | |

### (1) Fisher's exact test

#### 8.1.1.4. ORR vs HEMOGLOBIN

Table 7: HEMOGLOBIN by Overall response rate

| Hemoglobin (g/dL) | <10 (N=) | >=10 (N=) | Total (N=) | p-value |
|---|---|---|---|---|
| Overall Response Rate (confirmed) | | | | |
| N | | | | |
| No | | | | |
| Yes (CR/PR) | | | | |

### (1) Fisher's exact test

(\*) The percentages take into account missing data, the p-values do not

Table 8: HEMOGLOBIN by Overall response rate without UK/NE

| Hemoglobin (g/dL) | <10 (N=) | >=10 (N=) | Total (N=) | p-value |
|---|---|---|---|---|
| Overall Response Rate (confirmed) | | | | |
| N | | | | |
| Yes (CR/PR) | | | | |
| No | | | | |

### (1) Fisher's exact test

#### 8.1.1.5. ORR vs LIVER METASTASIS

Table 9: LIVER METASTASIS by Overall response rate

| Liver metastasis at baseline | No (N=) | Yes (N=) | Total (N=) | p-value |
|---|---|---|---|---|
| Overall Response Rate (confirmed) | | | | |
| N | | | | |
| No | | | | |
| Yes (CR/PR) | | | | |

### (1) Fisher's exact test

(\*) The percentages take into account missing data, the p-values do not

Table 10: LIVER METASTASIS by Overall response rate without UK/NE

| Liver metastasis at baseline | No (N=) | Yes (N=) | Total (N=) | p-value |
|---|---|---|---|---|
| Overall Response Rate (confirmed) | | | | |
| N | | | | |
| Yes (CR/PR) | | | | |
| No | | | | |

### (1) Fisher's exact test

### 8.2. SECONDARY OBJECTIVES

#### 8.2.1. TIME TO RESPONSE

To evaluate the time to response (TtR) associated with the study treatment, understood as the time from the first dose of the study treatment to the confirmed response (CR or PR) based on RECIST 1.1 criteria.

**Time to response (TtR)**: Time from first dosing date to the date of the documented ORR as determined using RECIST 1.1 criteria.

Table 55: Time to response

| Overall | Overall (N=) |
|------------------|--------------|
| Time to response | |
| (months) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |

#### 8.2.2. DURATION OF RESPONSE

**Duration of response (DoR)**: Time from first confirmed response (CR or PR) to the date of the documented PD as determined using RECIST 1.1 criteria or death due to any cause, whichever occurs first.

Table 56: Duration of response

| Overall | Overall (N=) |
|----------------------|--------------|
| Duration of response | |
| (months) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |

Table 57: Duration of response of responders (Best Overall Response CR or PR)

| Best Overall Response (Recist 1.1) | CR (N=) | PR (N=) | Total (N=) |
|--------------------------------------|---------|---------|------------|
| <b>Duration of response (months)</b> | | | |
| N | | | |
| Mean (95%CI) | | | |
| SD | | | |
| Median (95%CI) | | | |
| Range | | | |

Table 11: Patients with duration of response greater than 24 months

| Patient number | Hospital | Duration of response (months) | Best Overall Response<br>(Recist 1.1) |
|---|---|---|---|

Figure 5: Spider plot

### 8.2.3. CLINICAL BENEFIT RATE

To evaluate the clinical benefit rate (CBR), defined as the percentage of patients who have achieved complete response, partial response and stable disease. Stable disease should be maintained for at least 6 months to be considered as CBR event, from baseline (treatment start) to last tumor assessment with SD (or PR/CR in patients with non-confirmed response).

Table 58: Clinical benefit rate

| ClinicalBenefitRate | N | % | 95%CI |
|--------------------------|---|---|-------|
| No | | | |
| Yes (CR/PR/Manteined SD) | | | |
| Total | | | |

#### 8.2.4. FOLLOW-UP TIME

Table 59: Follow-up time in months (since study inclusion until death or last FU)

| Overall | Overall (N=) |
|----------------|--------------|
| Follow-up time | |
| (months) | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |

#### 8.2.5.PFS

Progression-free Survival (PFS): Median Progression free survival (mPFS) is defined as the time from the date of inclusion to the date of the first documented disease progression or death due to any cause, whichever occurs first. PFS will be determined based on tumour assessment (RECIST version 1.1 criteria). The local Investigator's assessments will be used for analyses. Patients who are alive and have not progressed at the last follow-up will be censored at the date of the last available image determination (CT scan or MRI). Patients with no additional image test other than that at baseline will be censored to the day after inclusion. Patients initiating new anticancer therapy (without progression to the study treatment) will be censored to the date of new anticancer therapy initiation.

Table 60: Progression information

| Progression | N | % | 95%CI |
|-------------|---|---|-------|
| No | | | |
| Yes | | | |
| Total | | | |

Table 61: Progression status

| Overall (N=) |
|--------------|

Figure 6: PFS

Table 62: Median/mean PFS (estimated by Kaplan-Meier)

| | Median (months) | CI 95% | RMST | CI 95% |
|---------------------------|-----------------|--------|------|--------|
| Progression Free Survival | | | | |

Table 63: PFS estimated survival ratio

| Progression Free<br>Survival | Events (%, total N) | Patients at risk | % estimated cumulative survival ratio | CI 95% |
|---|---|---|---|---|
| At 3 months | | | | |
| At 6 months | | | | |
| At 9 months | | | | |
| At 12 months | | | | |

#### 8.2.5.1. **PFS** vs AgE>70

Figure 7: PFS vs Age>70

Table 64: Median/mean PFS (estimated by Kaplan-Meier) vs Age>70

| | Median (months) | CI 95% | RMST | CI 95% |
|-----|-----------------|--------|------|--------|
| Yes | | | | |
| No | | | | |

Table 65: PFS estimated survival ratio vs Age>70

| PFS | Events (%, total N) | Patients at risk | % estimated cumulative survival ratio | CI 95% |
|---|---|---|---|---|
| Yes | | | | |
| At 3 months | | | | |
| At 6 months | | | | |
| At 9 months | | | | |
| At 12 months | | | | |
| No | | | | |
| At 3 months | | | | |
| At 6 months | | | | |
| At 9 months | | | | |
| At 12 months | | | | |

#### 8.2.5.2. PFS vs Renal Impairment

Figure 8: PFS vs Renal Impairment

Table 66: Median/mean PFS (estimated by Kaplan-Meier) vs Renal Impairment

| | Median (months) | CI 95% | RMST | CI 95% |
|-----|-----------------|--------|------|--------|
| Yes | | | | |
| No | | | | |

Table 67: PFS estimated survival ratio vs Renal Impairment

| PFS | Events (%, total N) | Patients at risk | % estimated cumulative survival ratio | CI 95% |
|---|---|---|---|---|
| Yes | | | | |
| At 3 months | | | | |
| At 6 months | | | | |
| At 9 months | | | | |
| At 12 months | | | | |
| No | | | | |
| At 3 months | | | | |
| At 6 months | | | | |
| At 9 months | | | | |
| At 12 months | | | | |

### 8.2.5.3. **PFS** vs **ECOG** 2

Figure 9: PFS vs ECOG 2

Table 68: Median/mean PFS (estimated by Kaplan-Meier) vs ECOG 2

| | Median (months) | CI 95% | RMST | CI 95% |
|-----|-----------------|--------|------|--------|
| Yes | | | | |
| No | | | | |

Table 69: PFS estimated survival ratio vs ECOG 2

| PFS | Events (%, total N) | Patients at risk | % estimated cumulative survival ratio | CI 95% |
|---|---|---|---|---|
| Yes | | | | |
| At 3 months | | | | |
| At 6 months | | | | |
| At 9 months | | | | |
| At 12 months | | | | |
| No | | | | |
| At 3 months | | | | |
| At 6 months | | | | |
| At 9 months | | | | |
| At 12 months | | | | |

### 8.2.5.4. PFS vs HEMOGLOBIN

Figure 10: PFS vs HEMOGLOBIN

Table 70: Median/mean PFS (estimated by Kaplan-Meier) vs HEMOGLOBIN

| | Median (months) | CI 95% | RMST | CI 95% |
|------|-----------------|--------|------|--------|
| <10 | | | | |
| >=10 | | | | |

Table 71: PFS estimated survival ratio vs HEMOGLOBIN

| PFS | Events (%, total N) | Patients at risk | % estimated cumulative survival ratio | CI 95% |
|---|---|---|---|---|
| <10 | | | | |
| At 3 months | | | | |
| At 6 months | | | | |
| At 9 months | | | | |
| At 12 months | | | | |
| >=10 | | | | |
| At 3 months | | | | |
| At 6 months | | | | |
| At 9 months | | | | |
| At 12 months | | | | |

#### 8.2.5.5. PFS vs LIVER METASTASIS

Figure 11: PFS vs LIVER METASTASIS

Table 72: Median/mean PFS (estimated by Kaplan-Meier) vs LIVER METASTASIS

| | Median (months) | CI 95% | RMST | CI 95% |
|-----|-----------------|--------|------|--------|
| No | | | | |
| Yes | | | | |

Table 73: PFS estimated survival ratio vs LIVER METASTASIS

| PFS | Events (%, total N) | Patients at risk | % estimated cumulative survival ratio | CI 95% |
|---|---|---|---|---|
| No | | | | |
| At 3 months | | | | |
| At 6 months | | | | |
| At 9 months | | | | |
| At 12 months | | | | |
| Yes | | | | |
| At 3 months | | | | |
| At 6 months | | | | |
| At 9 months | | | | |
| At 12 months | | | | |

### 8.2.6.OS

To determine the overall survival (OS) of patients with locally-advanced or mUC treated with the intended treatment regimen, understood as the time from first dosing date to the date of death. A subject who has not died will be censored at the last known date alive.

Table 74: Current situation information

| Status | N | % | 95%CI |
|--------|---|---|-------|
| Alive | | | |
| Death | | | |
| Total | | | |

Table 75: Death reason

| Overall | Overall (N=) |
|---------------------------------|--------------|
| Exitus Reason | |
| NA | |
| Progression disease | |
| Toxicity due to study treatment | |
| Other | |
| Exitus Reason Specify | |

Figure 12: OS

Table 76: Median/mean OS (estimated by Kaplan-Meier)

| | Median (months) | CI 95% | RMST | CI 95% |
|------------------|-----------------|--------|------|--------|
| Overall Survival | | | | |

Table 77: OS estimated survival ratio

| Overall<br>Survival | Events (%, total N) | Patients at risk | % estimated cumulative survival ratio | CI 95% |
|---|---|---|---|---|
| At 3 months | | | | |
| At 6 months | | | | |
| At 9 months | | | | |
| At 12 months | | | | |
| At 24 months | | | | |

#### 8.2.6.1. OS vs AgE>70

Figure 13: OS vs Age>70

Table 78: Median/mean OS (estimated by Kaplan-Meier) vs Age>70

| | Median (months) | CI 95% | RMST | CI 95% |
|-----|-----------------|--------|------|--------|
| Yes | | | | |
| No | | | | |

Table 79: OS estimated survival ratio vs Age>70

| os | Events (%, total N) | Patients at risk | % estimated cumulative survival ratio | CI 95% |
|---|---|---|---|---|
| Yes | | | | |
| At 3 months | | | | |
| At 6 months | | | | |
| At 9 months | | | | |
| At 12 months | | | | |
| No | | | | |
| At 3 months | | | | |
| At 6 months | | | | |
| At 9 months | | | | |
| At 12 months | | | | |

#### 8.2.6.2. OS VS RENAL IMPAIRMENT

Figure 14: OS vs Renal Impairment

Table 80: Median/mean OS (estimated by Kaplan-Meier) vs Renal Impairment

| | Median (months) | CI 95% | RMST | CI 95% |
|-----|-----------------|--------|------|--------|
| Yes | | | | |
| No | | | | |

Table 81: OS estimated survival ratio vs Renal Impairment

| os | Events (%, total N) | Patients at risk | % estimated cumulative survival ratio | CI 95% |
|---|---|---|---|---|
| Yes | | | | |
| At 3 months | | | | |
| At 6 months | | | | |
| At 9 months | | | | |
| At 12 months | | | | |

| os | Events (%, total N) | Patients at risk | % estimated cumulative survival ratio | CI 95% |
|---|---|---|---|---|
| No | | | | |
| At 3 months | | | | |
| At 6 months | | | | |
| At 9 months | | | | |
| At 12 months | | | | |

### 8.2.6.3. OS vs ECOG 2

Figure 15: OS vs ECOG 2

Table 82: Median/mean OS (estimated by Kaplan-Meier) vs ECOG 2

| | Median (months) | CI 95% | RMST | CI 95% |
|-----|-----------------|--------|------|--------|
| Yes | | | | |
| No | | | | |

Table 83: OS estimated survival ratio vs ECOG 2

| os | Events (%, total N) | Patients at risk | % estimated cumulative survival ratio | CI 95% |
|---|---|---|---|---|
| Yes | | | | |
| At 3 months | | | | |
| At 6 months | | | | |
| At 9 months | | | | |
| At 12 months | | | | |
| No | | | | |
| At 3 months | | | | |
| At 6 months | | | | |
| At 9 months | | | | |
| At 12 months | | | | |

### 8.2.6.4. OS vs HEMOGLOBIN

Figure 16: OS vs HEMOGLOBIN

Table 84: Median/mean OS (estimated by Kaplan-Meier) vs HEMOGLOBIN

| | Median (months) | CI 95% | RMST | CI 95% |
|------|-----------------|--------|------|--------|
| <10 | | | | |
| >=10 | | | | |

Table 85: OS estimated survival ratio vs HEMOGLOBIN

| os | Events (%, total N) | Patients at risk | % estimated cumulative survival ratio | CI 95% |
|---|---|---|---|---|
| <10 | | | | |
| At 3 months | | | | |
| At 6 months | | | | |
| At 9 months | | | | |
| At 12 months | | | | |
| >=10 | | | | |
| At 3 months | | | | |
| At 6 months | | | | |
| At 9 months | | | | |
| At 12 months | | | | |

#### 8.2.6.5. OS vs LIVER METASTASIS

Figure 17: OS vs LIVER METASTASIS

Table 86: Median/mean OS (estimated by Kaplan-Meier) vs LIVER METASTASIS

| | Median (months) | CI 95% | RMST | CI 95% |
|-----|-----------------|--------|------|--------|
| No | | | | |
| Yes | | | | |

Table 87: OS estimated survival ratio vs LIVER METASTASIS

| os | Events (%, total N) | Patients at risk | % estimated cumulative survival ratio | CI 95% |
|---|---|---|---|---|
| No | | | | |
| At 3 months | | | | |
| At 6 months | | | | |
| At 9 months | | | | |
| At 12 months | | | | |
| Yes | | | | |
| At 3 months | | | | |
| At 6 months | | | | |
| At 9 months | | | | |
| At 12 months | | | | |

# 9. SAFETY ANALYSIS

The following analyses in this section are carried out in the safety population (N = XX patients).

In the following tables, the adverse event which are not completely ruled out as toxicities or serious are considered toxicities and SAEs respectively.

Table 12: Overall safety

| Overall | Overall (N=) |
|----------------------------------------------|--------------|
| Adverse Events | - , |
| No | |
| Yes | |
| AE Grade >=3 | |
| No | |
| Yes | |
| Toxicity: AE related to Atezolizumab | |
| No | |
| Yes | |
| Toxicity: AE related to Cisplatin | |
| No | |
| Yes | |
| Toxicity: AE related to Gemcitabine | |
| No | |
| Yes | |
| Toxicity: AE related to all treatments | |
| No | |
| Yes | |
| Toxicity: AE related to any treatment | |
| No | |
| Yes | |
| Toxicity grade >=3 | |
| No | |
| Yes | |
| Toxicity related to Atezolizumab grade | |
| >=3 | |
| No | |
| Yes | |
| Toxicity related to Cisplatin grade >=3 | |
| No | |
| Yes | |
| Toxicity related to Gemcitabine grade | |
| >=3 | |
| No | |
| Yes | |
| Toxicity related to all treatments grade >=3 | |
| No<br>Voc | |
| Yes | |
| SAE<br>No. | |
| No | |

| Overall | Overall (N=) |
|---------|--------------|
| Yes | |

Table 13: Toxicities with 5% threshold

| Toxicity | Frequency | Percentage (%) |
|----------|-----------|----------------|

Table 14: Grade of toxicities with 5% threshold overall

| Toxicity | No | G-UK | G-1 | G-2 | G-3 | G-4 | G-5 |
|----------|----|------|-----|-----|-----|-----|-----|

Table 15: List of toxicities grade ≥ 3 in all patients

| Patient<br>Number | AE CTCAE | AE<br>Grade | AE<br>Related | AE Related to |
|-------------------|----------|-------------|---------------|---------------|

Table 16: AEs with 5% threshold

| AE | Frequency | Percentage (%) |
|----|-----------|----------------|

Table 17: Grade of AEs with 5% threshold overall

| AE | No | G-UK | G-1 | G-2 | G-3 | G-4 | G-5 |
|----|----|------|-----|-----|-----|-----|-----|

Table 18: List of all SAEs

| Patient | AE CTCAE | AE CTCAE | AE | AE Start | AE Stop | AE | AE Related | ΑE | AE |
|---|---|---|---|---|---|---|---|---|---|
| Number | AE CICAE | Other | Grade | Date | Date | Related | to | SAE | Intensity |

# 9.1. ANNEX 1

Table 19: List of all toxicities

| Patient<br>Number | AE CTCAE | AE CTCAE<br>Other | AE<br>Grade | AE Start<br>Date | AE Stop<br>Date | AE<br>Related | AE Related to | AE SAE Intensity |
|---|---|---|---|---|---|---|---|---|





Figure 20: Summary of adverse events.

All AEs have been grouped into blocks when the start date is consecutive to the end of the same previous AE (no more than 1 day has passed) for the same patient. The highest severity within the block is the one that remains. Additionally, if one of the events was related to the medication, that relationship is maintained for the entire block.

| | | SAE ( | No SAE (= Total<br>AEs - SAEs) | | | |
|---|---|---|---|---|---|---|
| Events | N pts<br>SAE | N<br>eventos<br>SAE | N<br>eventos<br>muerte | N SAE<br>Rit | N pts | N<br>eventos |

A threshold of 5% was set for No SAEs.